CLINICAL TRIAL: NCT01955525
Title: Long-term Follow-up of Health Related Quality of Life in Patients Hospitalised With Acute Coronary Syndrome: Evaluation of the Methods and Management of Acute Coronary Events (EMMACE)-3X
Brief Title: Long-term Follow-up of Health Related Quality of Life in Patients With Acute Coronary Syndrome
Acronym: EMMACE-3X
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Oras Alabas, Dr, University of Leeds
Other Study IDs: IRAS ID: 134080
Record Dates: First submitted 2013-09-28; First posted 2013-10-07 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; health related quality of life; mortality
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute coronary patients: Patients aged 18 and above who have been hospitalised with an ACS during the period of 2011 to 2013.

SUMMARY:
This study is aiming to i)measure longterm health related quality of life (HRQL) outcomes of the EMMACE3 patients hospitalised with acute coronary syndromes (ACS) and evaluate possible associations with their cardiovascular profile and to ii) Linkage these data to multiple electronic healthcare records

DETAILED DESCRIPTION:
Over the last few years the chance of dying from a heart attack in England and Wales has reduced dramatically. Even so, there remain huge differences in mortality between hospitals. For example, up to a third of patients with a heart attack who attend hospitals in England are more likely to die than would be expected. That is, the type of treatment and the risk of death depend upon where a patient lives and which hospital they attend. In part, the variation in death may be due to the services available at the hospital or to factors such as socioeconomic deprivation. It may also relate to other factors such as depression, cardiac rehabilitation, patient experience of hospital care and health quality of life.

Using statistical approaches that include measures of quality of life, we propose to examine data about heart attacks in England and investigate the 'postcode lottery of care'. This research is a long term followup that promote improved patient care. In doing so, different factors affecting cardiac rehabilitation will be highlighted and healthcare policy changed so that all patients will have an equal chance of surviving a heart attack.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18 years, both sexes, acute admission to hospital in England with an ACS, consented to participate in EMMACE3 study

Exclusion Criteria:

* Those in whom follow up would be inappropriate or impractical (for example patients in the terminal stages of an illness or requiring emergency treatment such that the gathering research data is not possible or appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been hospitalised with an ACS during the period of 2011 to 2013 and took part in EMMACE3 study(REC number 10/H1313/74)
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2013-11; Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | 10 years
  This research will therefore allow greater insights into the associations of patients and hospital characteristics with longerterm outcomes after ACS. It will identify good hospital practice and make recommendations for hospital care that will improve patient wellbeing.

SECONDARY OUTCOMES:
Mortality | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom